CLINICAL TRIAL: NCT01743586
Title: The Impact of Changes in Respiratory Muscle Function on Dyspnea, Functional Capacity, and Quality of Life in Patients With Advanced Lung Cancer & the Effects of Chest Physiotherapy Education Intervention
Brief Title: Respiratory Muscle Function Changes and Effects of Chest Physiotherapy Education Interventionin Advanced Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200912088R
Record Dates: First submitted 2010-03-16; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Chest physiotherapy; Respiratory muscle strength; Dyspnea, Functional capacity; Quality of life
MeSH Terms: conditions — Lung Neoplasms; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control (No Intervention)
  Interventions: Other: Chest physiotherapy education intervention

INTERVENTIONS:
Other: Chest physiotherapy education intervention — breathing exercise (diaphragmatic breathing and pursed-lip breathing cough training secretion mobilization (percussion and vibration) progressive muscle relaxation pacing and energy-saving techniques

SUMMARY:
The purpose for the 1st phase of this study are to exam longitudinal changes and the impact of various treatments on the respiratory muscle function, and the relations with dyspnea, functional capacity, quality of life, 6- and 12-month respiratory morbidity, and survival status (control group). The 2nd phase of this study will investigate the potential beneficial effects of chest physiotherapy in the same patient population (intervention group).

DETAILED DESCRIPTION:
Respiratory muscle function is critical for maintaining effective alveolar ventilation, and airway secretions clearance. The reduction in respiratory muscle function might lead to chronic respiratory insufficiency, and potentially to life-threatening problems. Respiratory muscle function and the impacts of various treatments regimens have not been investigated longitudinally in patients with advanced lung cancer patients.

The purposes for the 1st phase of this study are to exam longitudinal changes and the impact of various treatments on the respiratory muscle function, and the relations with dyspnea, functional capacity, quality of life, 6- and 12-month respiratory morbidity, and survival status (control group). The 2nd phase of this study will investigate the potential beneficial effects of chest physiotherapy in the same patient population (intervention group).

Methods: 102 patients with advanced lung cancer per group will be recruited from the National Taiwan University Hospital. Demographic and clinical signs/syndromes will be obtained from the chart. Pain and dyspnea will be measured using visual analog scale. Respiratory muscle strength will be tested by measuring maximal inspiratory and expiratory pressure (PImax and PEmax, respectively). Spirometric variables, forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) will be measured. Functional capacity will be measured using Karnofsky performance status and Simmonds functional assessment. Anxiety/depression symptom will be measured using Hospital Anxiety and Depression Scale. Quality of life will be measured using European Organization for Research and Treatment of Cancer, EORTC QLQ-C30 and LC13 questionnaire. Six- and 12-month respiratory complication morbidity and survival status will be recorded in the prospective nature.

Clinical relevance: The prevalence of lung cancer is increasing in the recent years. To understand the indications for chest physiotherapy (e.g., respiratory muscle weakness and its related sequels) and the effects of chest physiotherapy program will shed light on if routine chest physiotherapy should be implanted for patients with advanced lung cancer during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stage III/V lung cancer
* Normal cognition (a Mini Mental State Examination score of more than/equal to 24 points)
* Able to finish all tests

Exclusion Criteria:

* A clinical diagnosis affecting respiratory muscle function and functional activity performance (e.g. musculoskeletal disorders)
* Unable to perform acceptable-quality spirometry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Numbers of upper respiratory infections (URI) and respiratory infection related hospitalizations | 12 months after study entry
  Numbers of URIs and respiratory infection related hospitalizations were collected from out-patient and inpatient medical records.

SECONDARY OUTCOMES:
Funcional capacity Anxiety/depression symptom Quality of life Six- and 12-month respiratory complication morbidity and survival status | every 3 months up to 18 months post study entry
  Functional capacity measures included six-minute walk test, 50-foot walk with preferred and fast speed, and Barthel Index
Dyspnea and QoL | every 3 months up to 18 months
  Dyspnea was assessed using modified Borg scale and QoL was assessed using EORTC QLQ-C30 and LC13 questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, Ph.D., Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan